CLINICAL TRIAL: NCT03133676
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of KA34 Administered Via Intra-Articular Injection in Subjects With Osteoarthritis of the Knee
Brief Title: A Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of KA34 in Subjects With Knee Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calibr, a division of Scripps Research (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBR-KA34-3001
Record Dates: First submitted 2017-04-20; First posted 2017-04-28 (Actual); Results first posted 2021-05-17 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Arthritis; Joint Disease; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthritis; Joint Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KA34 Active Drug (Experimental): KA34 active drug in the dose range of 50 - 400 ug per knee
  Interventions: Drug: KA34
- Placebo (Placebo Comparator): Placebo is the formulation for KA34.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KA34 — 50 µg - 400 µg intra-articular injection (single or multiple doses)
  Other Names: KA-34
  Arms: KA34 Active Drug
Drug: Placebo — 50 µg - 400 µg intra-articular injection (single or multiple doses)
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and tolerability of KA34 when administered via intra-articular injection to subjects with osteoarthritis of the knee.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of KA34 when administered via intra-articular injection to subjects with osteoarthritis of the knee. OA patients are randomized to receive either placebo or KA34 active drug in the range of 50-400 ug by intra-articular injection. The first portion of the study is with single ascending doses, the second portion of the study is with multiple ascending doses.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of localized osteoarthritis of the knee
* Males willing to use contraception and females who are no longer able to bear children

Exclusion Criteria:

* Body Mass Index (BMI) > 40
* Grade 0, 3 or 4 osteoarthritis on the Kellgren and Lawrence classification system
* Injury to the knee or other joint within the last 12 months
* Receipt of any investigational product or experimental therapeutic procedure within the last 12 weeks

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lotz, MD, Study Director — Calibr, a division of Scripps Research
Locations (4):
- United States (4):
  - Diablo Clinical Research, Walnut Creek, California
  - Clinical Research of West Florida, Clearwater, Florida
  - Bioclinica Research, Orlando, Florida
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 subjects were randomized to 1 of 7 cohorts to receive KA34 or placebo. In the single-ascending dose (SAD) part, 24 subjects were randomized to receive a single dose of KA34 or placebo in 1 of 4 cohorts. After a thorough review of the Day 29 safety data from the SAD cohorts by the blinded Data Safety Monitoring Board, 36 subjects were randomized in the multiple-ascending dose (MAD) part of the study to receive 4 weekly doses of KA34 or placebo in 1 of 3 cohorts.
Pre-assignment Details: Subjects with a diagnosis of osteoarthritis (OA) of the knee as per the clinical and radiographic criteria of the American College of Rheumatology and joint pain with a visual analog scale score of ≥ 40 millimeters (mm) on a 100 mm scale on the index knee, determined by the Investigator at Screening were eligible to join the study.
Groups:
- Placebo (SAD): Subjects randomized to Cohorts 1 - 4 in the SAD part of the study received single intra-articular (IA) injections of matching placebo in the affected knee and were followed up until Day 29.
- Cohort 1: KA34 50 µg (SAD): Subjects received a single IA injection of 50 micrograms (µg) KA34 in the affected knee and were followed up until Day 29.
- Cohort 2: KA34 100 µg (SAD): Subjects received a single IA injection of 100 µg KA34 in the affected knee and were followed up until Day 29.
- Cohort 3: KA34 200 µg (SAD): Subjects received a single IA injection of 200 µg KA34 in the affected knee and were followed up until Day 29.
- Cohort 4: KA34 400 µg (SAD): Subjects received a single IA injection of 400 µg KA34 in the affected knee and were followed up until Day 29.
- Placebo (MAD): Subjects randomized to Cohorts 5 - 7 in the MAD part of the study received weekly IA injections of matching placebo in the affected knee for 4 weeks and were followed up until Day 180.
- Cohort 5: KA34 100 µg (MAD): Subjects received IA injections of 100 µg KA34 in the affected knee once weekly for 4 weeks and were followed up until Day 180.
- Cohort 6: KA34 200 µg (MAD): Subjects received IA injections of 200 µg KA34 in the affected knee once weekly for 4 weeks and were followed up until Day 180.
- Cohort 7: KA34 400 µg (MAD): Subjects received IA injections of 400 µg KA34 in the affected knee once weekly for 4 weeks and were followed up until Day 180.
Period: Overall Study
Arm/Group | Placebo (SAD) | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD) | Placebo (MAD) | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
Started | 6 | 3 | 3 | 6 | 6 | 9 | 9 | 9 | 9
Completed | 6 | 3 | 3 | 6 | 6 | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all subjects who received at least 1 dose of investigational product (IP) and were analyzed according to treatment received.
Groups:
- Placebo (SAD): Subjects randomized to Cohorts 1 - 4 in the SAD part of the study received single IA injections of matching placebo in the affected knee and were followed up until Day 29.
- Cohort 1: KA34 50 µg (SAD): Subjects received a single IA injection of 50 µg KA34 in the affected knee and were followed up until Day 29.
- Total: Total of all reporting groups
Arm/Group | Placebo (SAD) | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD) | Placebo (MAD) | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD) | Total
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 6 | 9 | 9 | 9 | 9 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 2 | 5 | 3 | 6 | 5 | 7 | 4 | 39
  >=65 years | 2 | 0 | 1 | 1 | 3 | 3 | 4 | 2 | 5 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 2 | 4 | 4 | 4 | 5 | 4 | 4 | 33
  Male | 1 | 2 | 1 | 2 | 2 | 5 | 4 | 5 | 5 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 4
  Not Hispanic or Latino | 6 | 3 | 3 | 6 | 6 | 9 | 7 | 9 | 7 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 2 | 1 | 4 | 1 | 2 | 0 | 11
  White | 6 | 3 | 1 | 4 | 4 | 5 | 8 | 6 | 9 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 3 | 6 | 6 | 9 | 9 | 9 | 9 | 60
Grade of Osteoarthritis (Kellgren and Lawrence radiological classification system) [Count of Participants; unit: Participants] — Grade 0: No radiographic features of OA present; Grade 1: Doubtful joint space narrowing (JSN) + possible osteophytic lipping; Grade 2: Definite osteophytes + possible JSN on anteroposterior weight-bearing radiograph; Grade 3: Multiple osteophytes, definite JSN, sclerosis, possible bony deformity; Grade 4: Large osteophytes, marked JSN, severe sclerosis + definite bony deformity;
  Participants
    Grade 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
    Grade 1 | 2 | 0 | 1 | 4 | 4 | 4 | 6 | 3 | 7 | 31
    Grade 2 | 4 | 1 | 2 | 2 | 2 | 5 | 3 | 6 | 2 | 27
    Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: SAD Part: Number of Subjects Who Experienced Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs were collected from time of first administration of IP (Day 1) until 28 days after the last administration of IP.
  The severity of TEAEs was classified by the investigator as mild, moderate or severe and graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The investigator also assessed relatedness of TEAEs. The number of subjects who experienced any TEAEs, serious TEAEs (SAE), related TEAEs and TEAEs with CTCAE Grade ≥ 3 are presented.
Time Frame: Day 1 up to Day 29
Population: The safety analysis set consisted of all subjects who received at least 1 dose of IP and were analyzed according to treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (SAD) | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD)
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 6
Participants
  At least 1 TEAE | 1 | 2 | 1 | 4 | 1
  At least 1 related TEAE | 0 | 0 | 0 | 2 | 0
  At least 1 severe TEAE | 0 | 0 | 0 | 0 | 0
  At least 1 severe related TEAE | 0 | 0 | 0 | 0 | 0
  At least 1 SAE | 0 | 0 | 0 | 1 | 0
  TEAE leading to discontinuation | 0 | 0 | 0 | 0 | 0
  TEAE leading to death | 0 | 0 | 0 | 0 | 0
  TEAE with CTCAE grade >=3 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: MAD Part: Number of Subjects Who Experienced TEAEs
Description: TEAEs were collected from time of first administration of IP (Day 1) until 30 days after the last administration of IP.
  The severity of TEAEs was classified by the investigator as mild, moderate or severe and graded using the CTCAE version 5.0. The investigator also assessed relatedness of TEAEs. The number of subjects who experienced any TEAEs, SAEs, related TEAEs and TEAEs with CTCAE Grade ≥ 3 are presented.
Time Frame: Day 1 up to Day 180
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (MAD) | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  At least 1 TEAE | 7 | 3 | 6 | 5
  At least 1 related TEAE | 4 | 1 | 1 | 0
  At least 1 severe TEAE | 1 | 0 | 0 | 0
  At least 1 severe related TEAE | 0 | 0 | 0 | 0
  At least 1 SAE | 0 | 0 | 0 | 0
  TEAE leading to discontinuation | 0 | 0 | 0 | 0
  TEAE leading to death | 0 | 0 | 0 | 0
  TEAE with CTCAE grade >=3 | 1 | 0 | 0 | 0

3. Secondary Outcome: SAD Part: Mean Change From Baseline in Hemoglobin at Day 8
Description: The mean changes from baseline at Day 8 in hemoglobin levels for subjects in the SAD part of the study are presented.
Time Frame: Baseline and Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams/deciliter (g/dL)
Arm/Group | Placebo (SAD) | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD)
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 6
grams/deciliter (g/dL) | -0.12 (0.58) | 0.77 (2.12) | -0.07 (0.81) | 0.08 (0.48) | -0.32 (0.50)

4. Secondary Outcome: MAD Part: Mean Change From Baseline in Hemoglobin at Day 180
Description: The mean changes from baseline at Day 180 in hemoglobin levels for subjects in the MAD part of the study are presented.
Time Frame: Baseline and Day 180
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo (MAD) | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
Number analyzed (Participants) | 9 | 9 | 9 | 9
g/dL | 0.36 (1.21) | -0.60 (1.01) | -0.48 (1.29) | -0.07 (0.19)

5. Secondary Outcome: SAD Part: Mean Change From Baseline in Hematocrit at Day 8
Description: The mean changes from baseline at Day 8 in hematocrit levels for subjects in the SAD part of the study are presented.
Time Frame: Baseline and Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: volume % of red blood cells (RBCs)
Arm/Group | Placebo (SAD) | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD)
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 6
volume % of red blood cells (RBCs) | -0.20 (1.61) | 2.40 (6.67) | -0.37 (2.70) | 0.12 (1.33) | -0.97 (1.58)

6. Secondary Outcome: MAD Part: Mean Change From Baseline in Hematocrit at Day 180
Description: The mean changes from baseline at Day 180 in hematocrit levels for subjects in the MAD part of the study are presented.
Time Frame: Baseline and Day 180
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: volume % of RBCs
Arm/Group | Placebo (MAD) | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
Number analyzed (Participants) | 9 | 9 | 9 | 9
volume % of RBCs | 42.68 (4.59) | 41.33 (4.77) | 42.12 (2.02) | 44.54 (2.35)

7. Secondary Outcome: SAD Part: Mean Change From Baseline in Total Bilirubin and Creatinine at Day 8
Description: The mean changes from baseline at Day 8 in total bilirubin and creatinine for subjects in the SAD part of the study are presented.
Time Frame: Baseline and Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams/dL (mg/dL)
Arm/Group | Placebo (SAD) | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD)
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 6
milligrams/dL (mg/dL)
  Total bilirubin | 0.023 (0.416) | 0.053 (0.137) | -0.033 (0.058) | 0.100 (0.179) | 0.037 (0.102)
  Creatinine | -0.038 (0.059) | 0.100 (0.200) | -0.063 (0.012) | -0.032 (0.041) | -0.117 (0.215)

8. Secondary Outcome: MAD Part: Mean Change From Baseline in Total Bilirubin and Creatinine at Day 180
Description: The mean changes from baseline at Day 180 in total bilirubin and creatinine for subjects in the MAD part of the study are presented.
Time Frame: Baseline and Day 180
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (MAD) | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
Number analyzed (Participants) | 9 | 9 | 9 | 9
mg/dL
  Total bilirubin | 0.067 (0.100) | -0.051 (0.153) | -0.017 (0.112) | -0.043 (0.264)
  Creatinine | -0.038 (0.100) | -0.006 (0.099) | 0.054 (0.112) | 0.030 (0.077)

9. Secondary Outcome: SAD Part: Mean Change From Baseline in Liver Enzymes at Day 8
Description: The mean changes from baseline at Day 8 in the following liver enzyme levels are presented for subjects in the SAD part of the study: alkaline phosphatase (ALP), alanine aminotransferase (ALT) and aspartate aminotransferase (AST).
Time Frame: Baseline and Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units/Liter (U/L)
Arm/Group | Placebo (SAD) | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD)
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 6
Units/Liter (U/L)
  ALP | 0.0 (3.8) | -7.7 (14.2) | 3.7 (7.0) | 0.0 (4.5) | 4.0 (11.7)
  ALT | 0.8 (4.5) | 3.7 (7.5) | -0.3 (1.5) | -1.3 (3.1) | -2.2 (4.3)
  AST | -0.2 (3.0) | 6.0 (10.1) | -2.7 (1.5) | -1.0 (2.5) | -1.2 (3.5)

10. Secondary Outcome: MAD Part: Mean Change From Baseline in Liver Enzymes at Day 180
Description: The mean changes from baseline at Day 180 in the following liver enzyme levels are presented for subjects in the MAD part of the study: ALP, ALT and AST.
Time Frame: Baseline and Day 180
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo (MAD) | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
Number analyzed (Participants) | 9 | 9 | 9 | 9
U/L
  ALP | -3.4 (8.8) | -0.2 (11.6) | -10.2 (13.8) | 1.1 (7.6)
  ALT | 2.1 (3.9) | -6.6 (21.1) | -3.8 (8.3) | 0.3 (3.3)
  AST | 0.7 (3.2) | -4.1 (12.8) | -1.1 (5.8) | -0.7 (3.1)

11. Secondary Outcome: SAD Part: Mean Change From Baseline in Systolic and Diastolic Blood Pressure at Day 8
Description: The mean changes from baseline at Day 8 in systolic blood pressure (SBP) and diastolic blood pressure (DBP) for subjects in the SAD part of the study are presented.
Time Frame: Baseline and Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters mercury (mmHg)
Arm/Group | Placebo (SAD) | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD)
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 6
millimeters mercury (mmHg)
  SBP | -7.3 (18.2) | 6.0 (12.2) | -11.3 (6.7) | 7.8 (10.9) | 3.7 (8.8)
  DBP | -2.0 (8.3) | 0.3 (10.6) | -8.3 (9.0) | 4.2 (9.2) | 9.0 (9.5)

12. Secondary Outcome: MAD Part: Mean Change From Baseline in SBP and DBP at Day 180
Description: The mean changes from baseline at Day 180 in SBP and DBP for subjects in the MAD part of the study are presented.
Time Frame: Baseline and Day 180
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo (MAD) | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
Number analyzed (Participants) | 9 | 9 | 9 | 9
mmHg
  SBP | 7.7 (13.3) | 8.9 (8.5) | -2.1 (15.3) | -0.3 (20.4)
  DBP | 6.6 (10.3) | 1.7 (8.5) | -3.0 (11.3) | 4.6 (9.4)

13. Secondary Outcome: SAD Part: Mean Change From Baseline in the QTcF Interval at Day 8
Description: The mean changes from baseline at Day 8 in the electrocardiogram (ECG) parameter QTcF interval for subjects in the SAD part of the study are presented.
Time Frame: Baseline and Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Placebo (SAD) | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD)
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 6
milliseconds (msec) | 2.3 (14.3) | 11.7 (6.8) | -3.7 (14.8) | -10.7 (25.3) | 3.5 (32.4)

14. Secondary Outcome: MAD Part: Mean Change From Baseline in the QTcF Interval at Day 180
Description: The mean changes from baseline at Day 180 in the ECG parameter QTcF interval for subjects in the MAD part of the study are presented.
Time Frame: Baseline and Day 180
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo (MAD) | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
Number analyzed (Participants) | 9 | 9 | 9 | 9
msec | 3.9 (13.5) | 1.9 (10.1) | -3.6 (14.7) | 3.4 (24.0)

15. Secondary Outcome: SAD Part: Number of Subjects With Injection Site TEAEs
Description: Physical examinations were conducted by a physician or another medically-qualified individual and findings were noted at the injection site during the study. The number of subjects with injection site TEAEs, including the following, are presented: Injection site erythema, Injection site hypersensitivity, Injection site inflammation, Injection site joint discomfort, Injection site joint inflammation, Injection site joint pain, Injection site joint swelling, Injection site nodule, Injection site pain and Injection site swelling.
Time Frame: Baseline up to Day 29
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (SAD) | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD)
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 6
Participants
  Injection site erythema | 0 | 0 | 0 | 1 | 0
  Injection site hypersensitvity | 0 | 0 | 0 | 0 | 1
  Injection site inflammation | 0 | 0 | 0 | 0 | 0
  Injection site joint discomfort | 0 | 0 | 0 | 0 | 0
  Injection site joint inflammation | 0 | 0 | 0 | 0 | 0
  Injection site joint pain | 0 | 0 | 0 | 0 | 0
  Injection site joint swelling | 0 | 0 | 0 | 0 | 0
  Injection site nodule | 0 | 0 | 0 | 0 | 0
  Injection site pain | 0 | 0 | 0 | 0 | 0
  Injection site swelling | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: MAD Part: Number of Subjects With Injection Site TEAEs
Description: as for outcome 15
Time Frame: Baseline up to Day 180
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (MAD) | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Injection site erythema | 0 | 0 | 0 | 0
  Injection site hypersensitivity | 0 | 0 | 0 | 0
  Injection site inflammation | 1 | 0 | 0 | 0
  Injection site joint discomfort | 1 | 1 | 1 | 1
  Injection site joint inflammation | 0 | 0 | 1 | 0
  Injection site joint pain | 2 | 0 | 2 | 1
  Injection site joint swelling | 2 | 0 | 0 | 0
  Injection site nodule | 1 | 0 | 0 | 0
  Injection site pain | 1 | 0 | 1 | 0
  Injection site swelling | 1 | 0 | 0 | 0

17. Secondary Outcome: SAD Part: Mean Maximum Plasma Concentration (Cmax)
Description: All Pharmacokinetic (PK) samples were analyzed by liquid chromatography with tandem mass spectrometry, using a validated, sensitive, specific method. Cmax values were obtained directly from the observed concentration versus time data, and the geometric mean Cmax values for subjects who received KA34 in the SAD part of the study are presented.
Time Frame: Pre-dose up to 4 hours post-dose on Day 1
Population: The PK analysis set consisted of all subjects who received KA34 and had at least 1 measured concentration at a scheduled PK time point after start of dosing without protocol violations or events with potential to affect the PK concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD)
Number analyzed (Participants) | 3 | 3 | 6 | 6
nanograms/milliliter (ng/mL) | 0.8528 (43.6) | 2.757 (29.9) | 5.732 (18.7) | 9.435 (41.4)

18. Secondary Outcome: MAD Part: Mean Cmax
Description: All PK samples were analyzed by liquid chromatography with tandem mass spectrometry, using a validated, sensitive, specific method. Cmax values were obtained directly from the observed concentration versus time data, and the geometric mean Cmax values for subjects who received KA34 in the MAD part of the study are presented.
Time Frame: Pre-dose up to 4 hours post-dose on Day 1 and pre-dose on Days 8, 15, 22 and 29
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
Number analyzed (Participants) | 9 | 9 | 9
ng/mL | 2.536 (33.7) | 4.807 (26.7) | 10.67 (40.3)

19. Secondary Outcome: SAD Part: Median Time to Maximum Observed Plasma Concentration (Tmax)
Description: All PK samples were analyzed by liquid chromatography with tandem mass spectrometry, using a validated, sensitive, specific method. Tmax was obtained directly from the observed concentration versus time data and the median Tmax values for subjects who received KA34 in the SAD part of the study are presented.
Time Frame: Pre-dose up to 4 hours post-dose on Day 1
Population: as for outcome 17
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD)
Number analyzed (Participants) | 3 | 3 | 6 | 6
hours (h) | 0.25 [0.25 to 0.52] | 0.50 [0.50 to 0.53] | 0.38 [0.22 to 0.53] | 0.30 [0.25 to 1.03]

20. Secondary Outcome: MAD Part: Median Tmax
Description: All PK samples were analyzed by liquid chromatography with tandem mass spectrometry, using a validated, sensitive, specific method. Tmax was obtained directly from the observed concentration versus time data and the median Tmax values for subjects who received KA34 in the MAD part of the study are presented.
Time Frame: Pre-dose up to 4 hours post-dose on Day 1 and pre-dose on Days 8, 15, 22 and 29
Population: as for outcome 17
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
Number analyzed (Participants) | 9 | 9 | 9
h | 0.50 [0.23 to 0.55] | 0.30 [0.25 to 0.50] | 0.50 [0.28 to 1.00]

21. Secondary Outcome: SAD Part: Mean Area Under the Concentration-time Curve From Time 0 to Time of Last Quantifiable Concentration (AUC[0-t])
Description: All PK samples were analyzed by liquid chromatography with tandem mass spectrometry, using a validated, sensitive, specific method. AUC(0-t) was calculated by linear up/log down trapezoidal summation, and the mean AUC(0-t) values for subjects who received KA34 in the SAD part of the study are presented.
Time Frame: Pre-dose up to 4 hours post-dose on Day 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD)
Number analyzed (Participants) | 3 | 3 | 6 | 6
ng*h/mL | 1.430 (0.2128) | 4.473 (2.555) | 9.933 (2.382) | 15.73 (2.515)

22. Secondary Outcome: MAD Part: Mean AUC(0-t)
Description: All PK samples were analyzed by liquid chromatography with tandem mass spectrometry, using a validated, sensitive, specific method. AUC(0-t) was calculated by linear up/log down trapezoidal summation, and the mean AUC(0-t) values for subjects who received KA34 in the MAD part of the study are presented.
Time Frame: Pre-dose up to 4 hours post-dose on Day 1 and pre-dose on Days 8, 15, 22 and 29
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
Number analyzed (Participants) | 9 | 9 | 9
ng*h/mL | 4.578 (1.312) | 7.077 (1.333) | 19.53 (9.554)

23. Secondary Outcome: SAD Part: Mean Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinite Time (AUC[0-inf])
Description: All PK samples were analyzed by liquid chromatography with tandem mass spectrometry, using a validated, sensitive, specific method. AUC(0-inf) was calculated by linear up/log down trapezoidal summation and extrapolated to infinity by the addition of the last quantifiable concentration (Clast) divided by the elimation rate constant (λz), i.e. AUC(0-t) + Clast/λz. The mean AUC(0-inf) values for subjects who received KA34 in the SAD part of the study are presented.
Time Frame: Pre-dose up to 4 hours post-dose on Day 1
Population: The PK analysis set consisted of all subjects who received KA34 and had at least 1 measured concentration at a scheduled PK time point after start of dosing without protocol violations or events with potential to affect the PK concentrations. Mean data is presented for subjects with data available for the parameter estimation.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD)
Number analyzed (Participants) | 2 | 2 | 6 | 5
ng*h/mL | 1.595 (0.2333) | 5.425 (3.953) | 11.09 (2.940) | 17.34 (3.626)

24. Secondary Outcome: MAD Part: Mean AUC(0-inf)
Description: All PK samples were analyzed by liquid chromatography with tandem mass spectrometry, using a validated, sensitive, specific method. AUC(0-inf) was calculated by linear up/log down trapezoidal summation and extrapolated to infinity by the addition of the last quantifiable concentration (Clast) divided by the elimation rate constant (λz), i.e. AUC(0-t) + Clast/λz. The mean AUC(0-inf) values are presented for subjects who received KA34 in the MAD part of the study.
Time Frame: Pre-dose up to 4 hours post-dose on Day 1 and pre-dose on Days 8, 15, 22 and 29
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
Number analyzed (Participants) | 9 | 8 | 9
ng*h/mL | 5.041 (1.556) | 7.370 (1.440) | 21.22 (11.05)

25. Secondary Outcome: SAD Part: Mean Apparent Terminal Half-life (t1/2)
Description: All PK samples were analyzed by liquid chromatography with tandem mass spectrometry, using a validated, sensitive, specific method. t1/2 was determined as the natural log of λz, i.e. as ln2/λz. Mean t1/2 values for subjects who received KA34 in the SAD part of the study are presented.
Time Frame: Pre-dose up to 4 hours post-dose on Day 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD)
Number analyzed (Participants) | 3 | 3 | 6 | 6
h | 1.253 (0.7117) | 1.420 (0.7072) | 1.145 (0.1666) | 1.222 (0.4439)

26. Secondary Outcome: MAD Part: Mean t1/2
Description: All PK samples were analyzed by liquid chromatography with tandem mass spectrometry, using a validated, sensitive, specific method. t1/2 was determined as the natural log of λz, i.e. as ln2/λz. Mean t1/2 values for subjects who received KA34 in the MAD part of the study are presented.
Time Frame: Pre-dose up to 4 hours post-dose on Day 1 and pre-dose on Days 8, 15, 22 and 29
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
Number analyzed (Participants) | 9 | 9 | 9
h | 1.072 (0.2567) | 0.9997 (0.2991) | 0.9286 (0.3044)

27. Secondary Outcome: SAD Part: Mean Apparent Clearance (CL/F)
Description: All PK samples were analyzed by liquid chromatography with tandem mass spectrometry, using a validated, sensitive, specific method. The CL/F after extravascular dosing was calculated as dose divided by AUC(0-inf), and is presented for subjects who received KA34 in the SAD part of the study.
Time Frame: Pre-dose up to 4 hours post-dose on Day 1
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD)
Number analyzed (Participants) | 2 | 2 | 6 | 5
L/h | 31.70 (4.667) | 25.10 (18.24) | 19.22 (5.466) | 23.92 (5.157)

28. Secondary Outcome: MAD Part: Mean CL/F
Description: All PK samples were analyzed by liquid chromatography with tandem mass spectrometry, using a validated, sensitive, specific method. The CL/F after extravascular dosing was calculated as dose divided by AUC(0-inf), and is presented for subjects who received KA34 in the MAD part of the study.
Time Frame: Pre-dose up to 4 hours post-dose on Day 1 and pre-dose on Days 8, 15, 22 and 29
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
Number analyzed (Participants) | 9 | 8 | 9
L/h | 21.43 (6.182) | 28.11 (5.695) | 23.85 (11.95)

29. Secondary Outcome: SAD Part: Mean Apparent Volume of Distribution (Vz/F)
Description: The Vz/F was calculated as dose divided by (λz*AUC[0-inf]), and the mean Vz/F values for subjects who received KA34 in the SAD part of the study are presented.
Time Frame: Pre-dose up to 4 hours post-dose on Day 1
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD)
Number analyzed (Participants) | 2 | 2 | 6 | 5
L | 38.25 (0.4950) | 34.30 (19.66) | 31.47 (9.479) | 35.56 (4.706)

30. Secondary Outcome: MAD Part: Mean Vz/F
Description: The Vz/F was calculated as dose divided by (λz*AUC[0-inf]), and the mean Vz/F values for subjects who received KA34 in the MAD part of the study are presented.
Time Frame: Pre-dose up to 4 hours post-dose on Day 1 and pre-dose on Days 8, 15, 22 and 29
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
Number analyzed (Participants) | 9 | 8 | 9
L | 32.51 (10.19) | 37.98 (13.46) | 30.00 (13.38)

ADVERSE EVENTS:
Time Frame: TEAEs were collected from time of first administration of IP (Day 1) up to 30 days after the last administration of IP (approximately 1 month for the SAD cohorts and approximately 6 months for the MAD cohorts).
Description: TEAEs are presented for the safety analysis set which consisted of all subjects who received at least 1 dose of IP and were analyzed according to treatment received.
Arm/Group | Placebo (SAD) | Cohort 1: KA34 50 µg (SAD) | Cohort 2: KA34 100 µg (SAD) | Cohort 3: KA34 200 µg (SAD) | Cohort 4: KA34 400 µg (SAD) | Placebo (MAD) | Cohort 5: KA34 100 µg (MAD) | Cohort 6: KA34 200 µg (MAD) | Cohort 7: KA34 400 µg (MAD)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/3 | 0/6 | 0/6 | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/3 | 1/6 | 0/6 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/6 | 2/3 | 1/3 | 4/6 | 1/6 | 7/9 | 3/9 | 6/9 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (SAD) (N=6) | Cohort 1: KA34 50 µg (SAD) (N=3) | Cohort 2: KA34 100 µg (SAD) (N=3) | Cohort 3: KA34 200 µg (SAD) (N=6) | Cohort 4: KA34 400 µg (SAD) (N=6) | Placebo (MAD) (N=9) | Cohort 5: KA34 100 µg (MAD) (N=9) | Cohort 6: KA34 200 µg (MAD) (N=9) | Cohort 7: KA34 400 µg (MAD) (N=9)
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (SAD) (N=6) | Cohort 1: KA34 50 µg (SAD) (N=3) | Cohort 2: KA34 100 µg (SAD) (N=3) | Cohort 3: KA34 200 µg (SAD) (N=6) | Cohort 4: KA34 400 µg (SAD) (N=6) | Placebo (MAD) (N=9) | Cohort 5: KA34 100 µg (MAD) (N=9) | Cohort 6: KA34 200 µg (MAD) (N=9) | Cohort 7: KA34 400 µg (MAD) (N=9)
Injection site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site hypersensitivity (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site joint discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Injection site joint pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site joint inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Injection site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site joint swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Injection site nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rabies (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT03133676/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT03133676/SAP_001.pdf